CLINICAL TRIAL: NCT06714955
Title: A Phase 1, Double-Blind, Parallel-arm, Placebo-Controlled, Multiple-dose Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of BGM0504 Injection Administered Subcutaneously in Non-diabetic Overweight or Obese Adult Subjects
Brief Title: Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of BGM0504 Injection in Non-diabetic Overweight or Obese Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BrightGene Bio-Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BGM0504-P1-001-US
Record Dates: First submitted 2024-11-27; First posted 2024-12-04 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2024-09

CONDITIONS: Non-diabetic Overweight or Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental: 10 mg BGM0504 10 milligrams (mg) BGM0504 administered subcutaneously (SC) once a week. (Experimental): Drug: BGM0504 Administered SC
  Interventions: Drug: Experimental: 10 mg BGM0504 10 milligrams (mg) BGM0504 administered subcutaneously (SC) once a week.
- Experimental: 15 mg BGM0504 15 mg BGM0504 administered SC once a week. (Experimental): Drug: BGM0504 Administered SC
  Interventions: Drug: Experimental: 15 mg BGM0504 15 mg BGM0504 administered SC once a week.
- Placebo Comparator: Placebo Placebo administered subcutaneously (SC) once a week. (Placebo Comparator): Drug: Placebo Administered SC
  Interventions: Drug: Placebo Comparator: Placebo Placebo administered subcutaneously (SC) once a week.

INTERVENTIONS:
Drug: Experimental: 10 mg BGM0504 10 milligrams (mg) BGM0504 administered subcutaneously (SC) once a week. — Drug: BGM0504 Administered SC
  Arms: Experimental: 10 mg BGM0504 10 milligrams (mg) BGM0504 administered subcutaneously (SC) once a week.
Drug: Experimental: 15 mg BGM0504 15 mg BGM0504 administered SC once a week. — Drug: BGM0504 Administered SC
  Arms: Experimental: 15 mg BGM0504 15 mg BGM0504 administered SC once a week.
Drug: Placebo Comparator: Placebo Placebo administered subcutaneously (SC) once a week. — Drug: Placebo Administered SC
  Arms: Placebo Comparator: Placebo Placebo administered subcutaneously (SC) once a week.

SUMMARY:
This is a Phase 1, double-blind, parallel-arm ,placebo-controlled study. The study will evaluate the pharmacokinetics (PK), pharmacodynamic (PD), safety and tolerability of BGM0504 following multiple subcutaneous (SC) administrations in non-diabetic overweight or obese adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) meeting one of the following requirements:

  1. Between ≥ 30.0 kg/m2 and ≤ 40.0 kg/m2 (obese); OR
  2. Between ≥ 27.0 kg/m2 and < 30.0 kg/m2 (overweight) with at least 1 of the following: 1) One or more of prediabetes (impaired fasting plasma glucose and/or abnormal glucose tolerance), grade 1 hypertension, simple fatty liver or dyslipidemia; 2) Weight-bearing joint pain; 3) Obesity causing dyspnea or obstructive sleep apnea syndrome
* Have a stable body weight (<5% self-reported change during the previous 8 weeks) before screening
* Capable of understanding the written informed consent document; willingly provides valid, signed written informed consent; willing and able to comply with the schedule, requirements and restrictions of the study.

Exclusion Criteria:

* Have allergic predisposition (allergic to 3 or more foods or drugs), or are allergic to glucagon-like peptide-1 (GLP-1) receptor agonists, or suffer from severe allergic diseases (asthma, urticaria, eczematous dermatitis).
* Have received GLP-1 receptor agonists or similar drugs containing the same target within 12 weeks before screening.
* Have received drugs that have an impact on body weight within 12 weeks before screening.
* Surgical treatment for obesity.
* Known type I/II diabetes.
* History of acute or chronic pancreatitis or pancreatic injury.
* History of drug abuse or alcoholism at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Number of treatment adverse events | 10 weeks
  The relationship of each adverse event tothe investigational product was assessed by the investigator

SECONDARY OUTCOMES:
Pharmacokinetic endpoint: Concentration of BGM0504 in plasma | 10 weeks
Change in fasting weight at week 10 | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron CPC, Inc, Baltimore, Maryland, United States